CLINICAL TRIAL: NCT03218839
Title: Evaluation of Safety, Efficacy and Acceptability of the PrePexTM Device for Rapid Scale-up of Adult Male Circumcision Programs in Zimbabwe, Phase III PrePexTM Field Implementation Trial With HIV Positive Adult Males
Brief Title: Evaluation of the PrePex Device for Rapid Scale-up of VMMC, Phase 3 Field Implementation Trial With HIV + Adult Males
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); Ministry of Health and Child Welfare, Zimbabwe (Other); University of Zimbabwe (Other); Zimbabwe Community Health Intervention Research Project (ZiCHIRe), Zimbabwe (Unknown)
Responsible Party: Principal Investigator, Scott Barnhart, Professor, Departments of Medicine and Global Health, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00000126
Record Dates: First submitted 2014-12-05; First posted 2017-07-17 (Actual); Last update posted 2017-07-17 (Actual); Status verified 2017-07

CONDITIONS: HIV Seropositivity
Keywords: PrePex; HIV Seropositivity
MeSH Terms: conditions — HIV Seropositivity

STUDY DESIGN:
Intervention Model Description: The study is a one arm, open label, prospective, cohort field study to assess the safety and acceptability of PrePex device circumcision device when performed by certified PrePex circumcision providers (physicians & nurses) in a HIV-infected male population.
Oversight: Data Monitoring Committee: No

ARMS (1):
- HIV+ PrePex (Experimental): PrePex male circumcision device
  Interventions: Device: PrePex male circumcision device

INTERVENTIONS:
Device: PrePex male circumcision device — PrePex non-surgical male circumcision device applied to eligible, consenting HIV-infected men in Zimbabwe to determine the rate of adverse events as compared to non HIV-infected men.

SUMMARY:
This study will assess the safety of the PrePex device as applied to HIV positive men by assessing the rate of clinical adverse events. The study will include adult, HIV + men who are eligible to receive the PrePex procedure per the Zimbabwe Ministry of Health and Child Care (MOHCC) eligibility criteria.

DETAILED DESCRIPTION:
According to mathematical modeling, Voluntary Medical Male Circumcision (VMMC) has the potential to have a major impact on reducing HIV incidence in areas with high HIV prevalence and low prevalence of male circumcision, as is the case in Zimbabwe. Male circumcision devices have the potential to accelerate VMMC scale-up as the procedure is faster and simpler and can be safely performed by nurses. However, fear of social stigma and desire to avoid HIV testing remain potential barriers to those HIV+ men who would otherwise seek out VMMC. Study subjects (n=400) are HIV+ males who elect to undergo VMMC with PrePex as a study subject, and healthcare workers involved in implementation of PrePex on HIV+ male subjects. The aim of the study is to determine if PrePex can be used safely among HIV+ men with similar rates of adverse events to HIV-uninfected men. If so, then the barrier of mandatory HIV testing as part of VMMC could be removed, encouraging more men to undergo the procedure. Determining PrePex safety in HIV+ men would also allow both those with unknown status and those with positive status to undergo MC with PrePex. Determining the barriers to performing VMMC among HIV+ men among healthcare workers, if any, would also inform future policy.

ELIGIBILITY:
Inclusion Criteria:

* Agrees to take an HIV test
* HIV sero-positive
* WHO HIV clinical stage 1 or 2
* Age 18 years and above
* Agrees to be circumcised by PrePex
* Able to understand the study procedures and requirements
* Completes VMMC counseling
* Agrees to return to the health care facility for follow-up visits or as instructed after this circumcision until complete healing 7 weeks from device application, or until cleared by a physician
* Able to comprehend and freely give informed consent for study participation

Exclusion Criteria:

* Known bleeding/coagulation abnormality (excessive bleeding from nosebleeds, pulled tooth, or gums)
* Uncontrolled diabetes (frequent treatment in a clinic or recent hospitalization for diabetes, frequent infections, hypertension, or kidney disease)
* Active genital infection, anatomic abnormality or any other condition, which in the opinion of the investigator prevents the subject from undergoing circumcision using PrePex.
* HIV sero-negative
* HIV status unknown
* WHO HIV stage 3 and above
* Does not agree to PrePex

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 430 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2016-02 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Rate of adverse events among HIV+ males using PrePex device | Device application through complete wound healing (up to 90 days)
  The primary safety endpoint is the incidence of clinical adverse events and device-related incidents.
  * Clinical related incidents such as the following:
    * Site bleeding (bleeding that cannot be stopped with pressure of 30 seconds and requires suturing)
    * Penis-wide diffuse hematoma
    * Penis-wide diffuse edema
    * Incision site infection and related symptoms
  * Device-related incidents
    * Necrotic Process not initiated
    * Device does not remain in situ for the full 7 days (displacement)
  Note: This list of AEs is not exhaustive.
  Severity of AE will be determined according to PEPFAR/OGAC guidelines

SECONDARY OUTCOMES:
Pain assessment at key time points | Placement through complete healing (up to 90 days)
  * Subject's subjective pain, tingling, and discomfort related to PrePex when applying the system, wearing it and removing it. This will be assessed by numeric pain, tingling and discomfort VAS scale (Pain = VAS x Duration in Minutes). Measured in the post placement recovery at 15 minutes after placement, and then 1, 2, and 3 hours post placement.
  * As the necrotic process initiates, it is expected that some of subjects will have temporary discomfort during the first 2 hours after deployment (hence anaesthetic cream), which vanishes thereafter for the rest of the weeklong period when the device is in place.
  * Some pain is expected for a short duration (about 10 seconds) when extracting the Inner Ring during the removal procedure.
Abstinence until complete wound healing | Post placement through complete healing (up to 90 days)
  Survival analysis of the timing of resumed sexual activity among subjects
Factors associated with abstinence until complete wound healing | Post placement through complete healing (approximately 90 days for men who participate in the qualitative component)
  Patient factors (knowledge, attitudes) associated with abstinence from sex until wound healing is complete
Time to complete healing | Device placement through complete healing (up to 90 days)
  Mean of days for complete healing (continuous measure) and factors associated with number of days to complete healing (continuous outcome - multiple linear regression)
  * A completely healed circumcision as defined as, "Intact epithelium (unbroken skin) covering the epithelial as judged by the provider on visual inspection, meaning that none of the following are present: sutures, scabbing, drainage, moisture, gaps between epithelial edges or ulceration.]
  * Optional validation by objective analysis of wounds by photographs
Cosmetic results | At complete healing (up to 90 days)
  * Objective analysis of photographs
  * Glans fully exposed (complete circumcision)
Patient satisfaction | 3 time points: Prior to the procedure, two weeks post-procedure, and 90 days post-procedure Device placement through ~90 days post procedure
  A composite measure created among patients involved in the qualitative component who will be asked about satisfaction with the PrePex™ MC procedure, barriers and motivators to uptake of VMMC through PrePex™, opinions around convenience of the device, tolerance of potential odour and whether participants would recommend PrePex™ MC to others.
Patient daily life | 3 time points: Prior to the procedure, two weeks post-procedure, and 90 days post-procedure Device placement through ~90 days post procedure
  Patients involved in the qualitative component will be asked about activities of daily living restrictions. They will complete a brief form that includes listing of activities of daily living, whether they are interrupted and for how long. This includes the average number of lost working hours (or potential working hours in unemployed). A composite measure will be created.
PrePex staff perceptions | 4 weeks after study implementation begins
  Responses by clinicians to Likert scale questions on their beliefs about PrePex VMMC and using this procedure on HIV+ men
PrePex staff clinical skills | At study closing,approximately 18 months after study initiation
  An overall assessment of clinician skills as a group will be made by combining and reporting on several indirect measures. Included measures will be the proportion of clients experiencing AEs and the average procedure time.
  • Assessing AE monitoring and reporting systems through
  * completeness of reporting
  * timeliness
PrePex AE monitoring and reporting systems | During all active follow-up: 90 days for participants
  An ongoing assessment of AE monitoring and reporting systems through
  * completeness of reporting
  * timeliness of reports
PrePex staff perceptions of their clinical skills | 4 weeks after study implementation begins
  Compilation report of Likert scale results from questions ascertaining PrepPex training, abilities, productivity and confidence.
PrePex staff satisfaction | 4 weeks after study implementation begins
  Compilation report on responses to likert scales question on their satisfaction performing PrePex on HIV+ men.

CONTACTS AND LOCATIONS:
Overall Officials: Scott Barnhart, MD, MPH, Principal Investigator — University of Washington
Locations (1):
- Zengeza Clinic, Chitungwiza, Harare, Zimbabwe